CLINICAL TRIAL: NCT01334879
Title: High Dose (2.0mg) Intravitreal Ranibizumab for Recalcitrant Radiation Retinopathy
Brief Title: High Dose Intravitreal Ranibizumab for Recalcitrant Radiation Retinopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The New York Eye Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Paul T. Finger, MD, Principal Investigator, The New York Eye Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FVF4981S
Record Dates: First submitted 2011-04-11; First posted 2011-04-13 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Radiation Retinopathy
Keywords: radiation; retinopathy; anti-VEGF; eye
MeSH Terms: conditions — Retinal Diseases | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With Loading Doses (Active Comparator): 5 patients will receive intravitreal injections every 30 days (+/- 7 days) for the first 4 months and every month thereafter until month 12 (maximum of 12 injections)
  Interventions: Drug: ranibizumab 2.0 mg
- Physician Discretion (Active Comparator): 5 patients will receive intravitreal ranibizumab every 30 days (+/- 7 days) on as needed basis based on the criteria defined in the study.
  Interventions: Drug: ranibizumab 2.0 mg

INTERVENTIONS:
Drug: ranibizumab 2.0 mg — Intravitreal ranibizumab (2.0 mg)
  Other Names: Lucentis

SUMMARY:
This study investigates the use of a high dose anti-VEGF agent for the treatment of radiation retinopathy in those patients who have recalcitrant disease.

DETAILED DESCRIPTION:
This study is an open-label, Phase I study of intravitreally administered ranibizumab in subjects with radiation retinopathy. This is a single center, non-randomized, active treatment study involving 10 consecutive patients. This study will evaluate the safety and tolerability of a high dose (2.0 mg) intravitreal ranibizumab and its effect on regression of radiation retinopathy and mean change in visual acuity.

ELIGIBILITY:
Inclusion Criteria

Subjects will be eligible if the following criteria are met:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 21 years
* History of a clinical diagnosis of radiation retinopathy
* Subjects who are at least 3 months and no more than 10 years from radiation therapy
* History of prior treatment for radiation retinopathy with incomplete response (eg. persistent edema, presence of hemorrhage, presence of exudates, etc
* ETDRS best corrected visual acuity of 20/400 or better in the study eye
* Ability to return for all study visits

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

* Pregnancy (positive pregnancy test) or lactation Premenopausal women not using adequate contraception. The following are considered effective means of contraception: surgical sterilization or use of oral contraceptives, barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel, an IUD, or contraceptive hormone implant or patch.
* Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
* Participation in another simultaneous medical investigation or trial
* Subject with significantly compromised visual acuity in the study eye due to concomitant ocular conditions.
* Subjects who have undergone intraocular surgery within last 60 days.
* Subjects who have had intravitreal anti-VEGF treatment within 30 days.
* Subjects who have had intravitreal triamcinolone acetonide within 4 months.
* Subjects who have had laser within 60 days.
* Inability to obtain photographs to document CNV (including difficulty with venous access).
* Subject with known adverse reaction to fluorescein dye.
* Subject has a history of any medical condition which would preclude scheduled visits or completion of study.
* Aphakia or absence of the posterior capsule in the study eye. Previous violation of the posterior capsule in the study eye is also excluded unless as a result of yttrium aluminum garnet (YAG) posterior capsulotomy in association with posterior chamber lens implantation..
* History of glaucoma filtering surgery in the study eye.
* Concurrent use of more than two therapies for glaucoma.
* Uncontrolled glaucoma in the study eye (defined as intraocular pressure >30 mm Hg despite treatment with anti-glaucoma medication)
* Inability to comply with study or follow-up procedure

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (allergy, infection, or change in vital signs) | Baseline, at day 7, then monthly
  All subjects will be assessed at baseline, at 7 days after first injection, and monthly for adverse events. The primary outcome measures for safety and tolerability are: 1. incidence and severity of ocular adverse events, as identified by eye examination (including best corrected visual acuity testing) and 2. Incidence and severity of other adverse events, as identified by physical examination, subject reporting, and changes in vital signs

SECONDARY OUTCOMES:
Number of participants with changes in central foveal thickness | Monthly, Report at Month 12
  This secondary outcome measure will evaluate the effect of ranibizumab in both groups (arms) on Regression of radiation retinopathy as measured by mean change in central retinal thickness as measured on optical coherence tomography (OCT) compared to baseline
Number of participants with changes in visual acuity | Monthly, Report at Month 12
  Each month each subject will be tested for best corrected visual acuity as compared to baseline.
Number of injections each group (arm) has received | Monthly, Report at Month 12
  Each group (arm) will be assessed for the number of monthyl injections received through Month 12.
Number of participants with qualitative changes in retinopathy on ophthalmoscopy and fluorescein angiography | Monthly Report at Month 12
  Evaluation of both arms on qualitative change in exudates, retinal hemorrhage, microaneurym and neovascularization) as seen on ophthalmoscopy/color photography and fluorescein angiography compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Paul T Finger, MD, Principal Investigator — The New York Eye Cancer Center
Locations (1):
- The New York Eye Cancer Center, New York, New York, United States

REFERENCES:
- See also: Dr. Finger's Radiation Retinopathy Studies — http://www.ncbi.nlm.nih.gov/pubmed?term=radiation%20retinopathy%20Finger%20PT